CLINICAL TRIAL: NCT04198298
Title: Prospective Comparative Randomized Clinical Trial of Three Endodontic Retrograde Filling Materials
Brief Title: Prospective Clinical Trial of Three Apical Sealing Materials
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of the Pacific (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-60
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Periapical Abscess
Keywords: Cone-Beam Computed Tomography; Microsurgery; Bone Regeneration; Biocompatible Materials
MeSH Terms: conditions — Periapical Abscess | interventions — EndoSequence root repair material; ProRoot MTA; tricalcium silicate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 EndoSequence (Active Comparator): The EndoSequence® retrograde sealing material was used to provide a biologic seal at the apex.
  Interventions: Drug: EndoSequence
- Group 2 ProRoot MTA (Active Comparator): The ProRoot® MTA retrograde sealing material was used to provide a biologic seal at the apex.
  Interventions: Drug: ProRoot MTA
- Group 3 Biodentine (Active Comparator): The Biodentine® retrograde sealing material was used to provide a biologic seal at the apex.
  Interventions: Drug: Biodentine

INTERVENTIONS:
Drug: EndoSequence — The EndoSequence® retrograde sealing material was used to provide a biologic seal at the apex.
  Other Names: EndoSequence®
  Arms: Group 1 EndoSequence
Drug: ProRoot MTA — The ProRoot® MTA retrograde sealing material was used to provide a biologic seal at the apex.
  Other Names: ProRoot® MTA
  Arms: Group 2 ProRoot MTA
Drug: Biodentine — The Biodentine® retrograde sealing material was used to provide a biologic seal at the apex.
  Other Names: Biodentine®
  Arms: Group 3 Biodentine

SUMMARY:
This prospective comparative randomized clinical trial compares healing and bony regeneration in patients who received 1 of 3 different retrograde filling materials following microsurgical apicoectomies for the treatment of periapical lesions of endodontic origin.

DETAILED DESCRIPTION:
A prospective comparative randomized clinical trial was designed to evaluate the healing and bony regeneration in patients who received 1 of 3 different retrograde filling materials (EndoSequence®, ProRoot® MTA, or Biodentine®) following microsurgical apicoectomies for the treatment of periapical lesions of endodontic origin.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, American Society of Anesthesiologists (ASA) classification I and II
* Any tooth with a single chronic periapical lesion requiring apical microsurgery
* Informed consent signed prior to surgery

Exclusion Criteria:

* Background of drug/alcohol abuse
* Adjacent periapical lesion
* Periodontal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-11-02 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Rate of remineralization | 6 months
  The pace at which new bone is redeposited